CLINICAL TRIAL: NCT01836523
Title: The Efficacy and Safety of Liraglutide as Adjunct Therapy to Insulin in the Treatment of Type 1 Diabetes. A 52-week Randomised, Treat-to-target, Placebo-controlled, Double Blinded, Parallel Group, Multinational, Multi-centre Trial
Brief Title: The Efficacy and Safety of Liraglutide as Adjunct Therapy to Insulin in the Treatment of Type 1 Diabetes
Acronym: ADJUNCT ONE™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9211-3919; 2012-003580-21 (EudraCT Number); U1111-1133-0590 (Other: WHO)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Liraglutide 0.6 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 1.2 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 1.8 mg + insulin (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide placebo 0.6 mg + insulin (Placebo Comparator)
  Interventions: Drug: placebo
- Liraglutide placebo 1.2 mg + insulin (Placebo Comparator)
  Interventions: Drug: placebo
- Liraglutide placebo 1.8 mg + insulin (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 0.6 mg + insulin
Drug: placebo — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 0.6 mg + insulin
Drug: liraglutide — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 1.2 mg + insulin
Drug: placebo — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 1.2 mg + insulin
Drug: liraglutide — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide 1.8 mg + insulin
Drug: placebo — Subjects randomised to 0.6 mg liraglutide treatment or liraglutide placebo as an add-on to their pre-trial insulin treatment will remain on this dose throughout the study (52 weeks). Administered subcutaneously (s.c., under the skin) once daily.
  Arms: Liraglutide placebo 1.8 mg + insulin

SUMMARY:
This trial is conducted globally. The aim of the trial is to confirm the efficacy and safety of liraglutide as adjunct therapy to insulin in the treatment of type 1 diabetes. The total trial duration per subject is approximately 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* - Informed consent obtained
* - Type 1 diabetes mellitus for 12 months or longer
* - Basal bolus or CSII (Continuous Subcutaneous Insulin Infusion, insulin pump) treatment for 6 months or longer
* - Stable insulin treatment for the last 3 months prior to Screening, as judged and documented by the investigator
* - HbA1c 7.0-10% (Diabetes Control and Complications Trial (DCCT)), both inclusive, (corresponding to 53-86 mmol/mol (International Federation of Clinical Chemistry (IFCC))
* - Ability and willingness to comply with all protocol procedures e.g. correct handling of trial product, complete trial related questionnaires, diaries, self-monitoring of plasma glucose, self titration of insulin and attend all scheduled visits

Exclusion Criteria:

* - Prior use of glucagon-like peptide-1 (GLP-1) receptor agonist or dipeptidyl peptidase IV (DPP-4) inhibitors
* - Use of any medication, which in the investigator's opinion could interfere with the glycaemic control or affect the subject's safety.Premix insulin is not allowed
* - Known proliferative retinopathy or maculopathy requiring acute treatment
* - Severe neuropathy, in particular autonomic neuropathy, i.e. gastroparesis, as judged by the investigator
* - Uncontrolled/ untreated blood pressure at screening above 160 mmHg for systolic or above 100 mmHg for diastolic
* - History of acute or chronic pancreatitis
* - Screening calcitonin value equal to or above 50 ng/L
* - Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia type 2 (MEN2)
* - Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (160):
- United States (63):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Metarie, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Springfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Upper Darby, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Summerville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, El Paso, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Bennington, Vermont
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Federal Way, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Argentina (5):
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mendoza
  - Novo Nordisk Investigational Site, Morón
- Australia (5):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Elizabeth Vale, South Australia
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Melbourne, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Belgium (4):
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Canada (12):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Barrie, Ontario
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Oakville, Ontario
  - Novo Nordisk Investigational Site, Thornhill, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
- Finland (5):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Seinäjoki
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (13):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Poitiers
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Saint-Priest-en-Jarez
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (9):
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Israel (5):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
- Netherlands (7):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Leiden
  - Novo Nordisk Investigational Site, Nijmegen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Venlo
- Norway (5):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Gjettum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Stavanger
- Poland (4):
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Puławy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Russia (4):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Volgograd
- Sweden (3):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- Ukraine (4):
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Poltava
  - Novo Nordisk Investigational Site, Zhytomyr
- United Kingdom (10):
  - Novo Nordisk Investigational Site, Blackburn
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Durham
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Southall
  - Novo Nordisk Investigational Site, St Helens
  - Novo Nordisk Investigational Site, Stevenage

REFERENCES:
- [Result] Mathieu C, Zinman B, Hemmingsson JU, Woo V, Colman P, Christiansen E, Linder M, Bode B; ADJUNCT ONE Investigators. Efficacy and Safety of Liraglutide Added to Insulin Treatment in Type 1 Diabetes: The ADJUNCT ONE Treat-To-Target Randomized Trial. Diabetes Care. 2016 Oct;39(10):1702-10. doi: 10.2337/dc16-0691. Epub 2016 Aug 9. PMID 27506222
- [Derived] Shah VN, Agesen RM, Bardtrum L, Christiansen E, Snaith J, Greenfield JR. Determinants of Liraglutide Treatment Discontinuation in Type 1 Diabetes: A Post Hoc Analysis of ADJUNCT ONE and ADJUNCT TWO Randomized Placebo-Controlled Clinical Studies. J Diabetes Sci Technol. 2025 Mar;19(2):321-331. doi: 10.1177/19322968241305647. Epub 2024 Dec 24. PMID 39717993
- [Derived] Dejgaard TF, von Scholten BJ, Christiansen E, Kreiner FF, Bardtrum L, von Herrath M, Mathieu C, Madsbad S; ADJUNCT ONE and ADJUNCT TWO Investigators. Efficacy and safety of liraglutide in type 1 diabetes by baseline characteristics in the ADJUNCT ONE and ADJUNCT TWO randomized controlled trials. Diabetes Obes Metab. 2021 Dec;23(12):2752-2762. doi: 10.1111/dom.14532. Epub 2021 Sep 28. PMID 34463425
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 177 sites in 17 countries: Argentina: 6, Australia: 5, Belgium: 4, Canada: 14, Germany: 8, Finland: 6, France: 13, United Kingdom: 10, Ireland: 5, Israel: 6, Netherlands: 6, Norway: 5, Poland: 5, Russia: 5, Sweden: 4, Ukraine: 5, United States: 70
Pre-assignment Details: Eligible subjects were randomised in a 3:3:3:1:1:1 manner to receive liraglutide (0.6 mg, 1.2 mg or 1.8 mg) or placebo (0.1 mL, 0.2 mL or 0.3 mL), both adjunct to insulin treatment.
Groups:
- Liraglutide 0.6 mg: Subjects received liraglutide 0.6 mg once daily (OD) subcutaneously for 52 weeks in addition to their pre-trial insulin treatment.
- Liraglutide 1.2 mg: Subjects received liraglutide 0.6 mg OD subcutaneously for 2 weeks followed by 1.2 mg OD subcutaneously up to week 52 in addition to their pre-trial insulin treatment.
- Liraglutide 1.8 mg: Liraglutide 0.6 mg OD subcutaneously for 2 weeks followed by 1.2 mg OD subcutaneously for 2 weeks (weeks 2-4) followed by 1.8 mg OD subcutaneously up to week 52 in addition to their pre-trial insulin treatment.
- Placebo: Subjects received placebo (matched to liraglutide 0.6, 1.2 and 1.8 mg) OD subcutaneously as an add-on to their pre-trial insulin treatment. Placebo 0.1 mL (placebo matched to liraglutide 0.6 mg): Subjects received 0.1 mL liraglutide placebo for 52 weeks. Placebo 0.2 mL (placebo matched to liraglutide 1.2 mg): Subjects received 0.1 mL for 2 weeks followed by 0.2 mL up to week 52. Placebo 0.3 mL (placebo matched to liraglutide 1.8 mg): Subjects received 0.1 mL for 2 weeks followed by 0.2 mL for next 2 weeks and 0.3 mL up to week 52. All the 3 placebo doses were pooled for data analysis.
Period: Overall Study
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Started | 351 | 350 | 349 | 348
Exposed | 350 | 348 | 347 | 348
Completed | 300 | 265 | 258 | 274
Not Completed | 51 | 85 | 91 | 74
Not completed — Adverse Event | 15 | 41 | 49 | 14
Not completed — Protocol Violation | 6 | 3 | 2 | 4
Not completed — Met Withdrawal Criteria | 13 | 13 | 21 | 27
Not completed — Unclassified | 17 | 28 | 19 | 29

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose and had any post-randomisation data. Five subjects, who started the study, were excluded because of no exposure to study drug and 4 subjects were excluded because of non-availability of post-baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo | Total
Number analyzed (Participants) | 350 | 346 | 346 | 347 | 1389
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.78) | 43.9 (13.06) | 43.7 (13.33) | 43.4 (12.57) | 43.7 (12.93)
Gender [Count of Participants; unit: Participants]
  Female | 186 | 179 | 181 | 180 | 726
  Male | 164 | 167 | 165 | 167 | 663
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.18 (0.738) | 8.16 (0.779) | 8.14 (0.740) | 8.15 (0.728) | 8.16 (0.746)
Body weight [Mean (Standard Deviation); unit: kg] | 86.54 (17.338) | 85.39 (17.210) | 86.27 (17.321) | 86.41 (17.768) | 86.15 (17.397)
Total daily actual insulin dose-continuous subcutaneous insulin infusion [Geometric Mean (Full Range); unit: units] — Total insulin daily dose of subjects who were on continuous subcutaneous insulin infusion treatment. Number of subjects analysed=69 (liraglutide 0.6 mg), 99 (liraglutide 1.2 mg), 113 (liraglutide 1.8 mg), 95 (Placebo).
  units | 52.97 [13.8 to 137.1] | 50.73 [19.7 to 160.5] | 50.46 [8.7 to 150.2] | 49.18 [3.9 to 176.1] | 50.65 [3.9 to 176.1]
Total daily actual insulin dose - Multiple daily injections [Geometric Mean (Full Range); unit: units] — Total insulin daily dose of subjects who were on multiple daily insulin injection treatment. Number of subjects analysed=277 (liraglutide 0.6 mg), 242 (liraglutide 1.2 mg), 227 (liraglutide 1.8 mg), 250 (Placebo).
  units | 59.54 [22.9 to 181.6] | 59.61 [16 to 282.5] | 62.52 [16.4 to 271.3] | 62.42 [20.3 to 230] | 60.94 [16 to 282.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c at week 52. Missing values were handled by using a mixed model for repeated measurements (MMRM).
Time Frame: Week 0, week 52
Population: Full analysis set. Number of subjects analysed=subjects with any post-baseline HbA1c data.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 334 | 312 | 305 | 324
percentage of glycosylated haemoglobin | -0.45 (0.741) | -0.50 (0.767) | -0.54 (0.729) | -0.34 (0.707)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; Analysis was performed using MMRMs where all post-baseline measurements for the specific variable from planned visits up to week 52 and obtained no later than 1 day after withdrawal from treatment were entered as the dependent variable, and visit, treatment, country and the stratification variable (4 levels: HbA1c < 8.5% and ≥8.5%, each intersected by BMI≤27 kg/m2 and >27 kg/m2) were included as fixed factors and the corresponding baseline value as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper bound of 95% confidence interval was <0.3; Treatment difference = -0.20, 95% CI 2-sided [-0.32 to -0.07]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper bound of 95% confidence interval was <0.3; Treatment difference = -0.15, 95% CI 2-sided [-0.27 to -0.03]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper bound of 95% confidence interval was <0.3; Treatment difference = -0.09, 95% CI 2-sided [-0.21 to 0.03]

2. Primary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight at week 52. Missing values were handled by using a MMRM.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of subjects analysed=subjects with any post-baseline body weight data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 324 | 300 | 298 | 311
kg | -1.34 (4.183) | -2.73 (4.524) | -4.02 (4.873) | 0.94 (3.828)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -4.90, 95% CI 2-sided [-5.65 to -4.16]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -3.55, 95% CI 2-sided [-4.29 to -2.81]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -2.19, 95% CI 2-sided [-2.91 to -1.47]

3. Primary Outcome: Change From Baseline in Total Daily Insulin Dose
Description: Change from baseline in total daily insulin dose at week 52. Change from baseline was represented in terms of ratio to baseline for insulin dose i.e. Total daily insulin dose at week 52/total daily insulin dose at baseline. Missing values were handled by using a MMRM.
Time Frame: Week 0, week 52
Population: Full analysis set. Number of subjects analysed=subjects with any post-baseline total insulin daily dose data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 337 | 328 | 331 | 341
ratio | 1.04 (23.75) | 0.98 (26.66) | 0.95 (24.21) | 1.04 (26.69)
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; Analysis was done using MMRMs where all post-baseline measurements for specific variable from planned visits up to week 52 and obtained no later than 1 day after withdrawal from treatment were entered as dependent variable, and visit, treatment, country and stratification variable (4 levels: HbA1c < 8.5% and ≥8.5%, each intersected by BMI≤27 kg/m2 and >27 kg/m2) were included as fixed factors and the corresponding baseline value as covariate. The measurements were log-transformed before analysis; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment ratio = 0.92, 95% CI 2-sided [0.88 to 0.96]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0148, Mixed Models Analysis; Treatment ratio = 0.95, 95% CI 2-sided [0.91 to 0.99]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9615, Mixed Models Analysis; Treatment ratio = 1.00, 95% CI 2-sided [0.96 to 1.04]

4. Secondary Outcome: Number of Treatment-emergent Symptomatic Hypoglycaemic Episodes
Description: This is a confirmatory secondary endpoint. Symptomatic hypoglycaemic episodes were defined as: 1) Severe according to the American Diabetes Association (ADA) classification: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. OR 2) Self-monitoring of plasma glucose value of <3.1 mmol/L, with symptoms consistent with hypoglycaemia. A treatment emergent episode is defined as an episode with onset date (or increase in severity) on or after first day of exposure to randomised treatment and up to last dose + 7 days.
Time Frame: Weeks 0-52
Population: The safety analysis set included all randomised subjects exposed to at least one dose of liraglutide or placebo.
Measure: Number; unit: episodes
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Number analyzed (Participants) | 350 | 348 | 347 | 348
episodes | 4954 | 4602 | 4614 | 3654
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Placebo; The endpoint was analysed using a negative binomial regression model with a log-link function and the log of the time period in which an occurrence of a hypoglycaemic episode was considered treatment emergent as offset. The model included fixed factors (treatment, country, stratification group) and a covariate (baseline HbA1c); Test type: Superiority or Other; p = 0.0081, Negative binomial regression; Rate ratio = 1.31, 95% CI 2-sided [1.07 to 1.59]
Statistical Analysis 2: Comparison: Liraglutide 1.2 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0219, Negative binomial regression; Rate ratio = 1.27, 95% CI 2-sided [1.03 to 1.55]
Statistical Analysis 3: Comparison: Liraglutide 0.6 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1079, Negative binomial regression; Rate ratio = 1.17, 95% CI 2-sided [0.97 to 1.43]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: A treatment emergent adverse event is defined as an event with onset date (or increase in severity) on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Arm/Group | Liraglutide 0.6 mg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 35/350 | 36/348 | 29/347 | 38/348
Other Adverse Events (participants affected / at risk) | 259/350 | 263/348 | 282/347 | 224/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.6 mg (N=350) | Liraglutide 1.2 mg (N=348) | Liraglutide 1.8 mg (N=347) | Placebo (N=348)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melkersson-Rosenthal syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biopsy prostate (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 3 (4) | 3 (4) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 7 (8) | 5 (5) | 13 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 5 (5) | 3 (3) | 6 (7) | 6 (7)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Popliteal artery entrapment syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.6 mg (N=350) | Liraglutide 1.2 mg (N=348) | Liraglutide 1.8 mg (N=347) | Placebo (N=348)
Abdominal pain (Gastrointestinal disorders) | 20 (32) | 16 (20) | 29 (41) | 8 (9)
Constipation (Gastrointestinal disorders) | 17 (20) | 28 (30) | 26 (28) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 41 (52) | 50 (69) | 64 (92) | 38 (50)
Dyspepsia (Gastrointestinal disorders) | 26 (37) | 27 (41) | 38 (48) | 8 (8)
Nausea (Gastrointestinal disorders) | 112 (146) | 141 (196) | 172 (271) | 42 (52)
Vomiting (Gastrointestinal disorders) | 24 (26) | 44 (58) | 64 (106) | 21 (26)
Fatigue (General disorders) | 17 (18) | 22 (24) | 18 (21) | 16 (18)
Gastroenteritis (Infections and infestations) | 21 (25) | 15 (17) | 29 (32) | 15 (21)
Gastroenteritis viral (Infections and infestations) | 12 (14) | 6 (6) | 18 (24) | 8 (10)
Influenza (Infections and infestations) | 29 (32) | 17 (26) | 25 (28) | 24 (30)
Nasopharyngitis (Infections and infestations) | 105 (175) | 81 (124) | 83 (145) | 85 (130)
Sinusitis (Infections and infestations) | 24 (35) | 17 (22) | 16 (21) | 21 (31)
Upper respiratory tract infection (Infections and infestations) | 33 (37) | 23 (37) | 43 (59) | 40 (58)
Urinary tract infection (Infections and infestations) | 18 (28) | 14 (21) | 20 (26) | 11 (15)
Decreased appetite (Metabolism and nutrition disorders) | 31 (32) | 43 (45) | 64 (70) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (29) | 17 (26) | 22 (38) | 17 (28)
Hypoglycaemia (Metabolism and nutrition disorders) | 26 (32) | 13 (18) | 20 (37) | 24 (35)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 22 (24) | 18 (19) | 16 (16)
Headache (Nervous system disorders) | 56 (78) | 46 (85) | 49 (119) | 40 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 7 (8) | 10 (12) | 21 (24)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 22 (24) | 28 (32) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk commits to communicating, and otherwise making available for public disclosure, results of trials regardless of outcome.At the end of the trial, one or more public disclosures may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.